CLINICAL TRIAL: NCT07305389
Title: The MUSICare Project: Effects of Differentiated Music Exposure on Exercise-Related Affect Among Cardiac Rehabilitation Inpatients
Acronym: MUSICare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elena Tessitore (Other)
Responsible Party: Sponsor-Investigator, Elena Tessitore, MD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0424; SNCTP000006164 (Other: HumRes)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Rehabilitation Exercise
Keywords: cardiac rehabilitation; music; physical activity; affective valence
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with repeated-measures and crossover design with full counterbalancing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MFH (Experimental): Music in the First Half of the Exercise Session
  Interventions: Other: Music listening during physical exercise
- MSH (Experimental): Music in the Second Half of the Exercise Session
  Interventions: Other: Music listening during physical exercise
- MT (Experimental): Music Throughout the Exercise Session
  Interventions: Other: Music listening during physical exercise
- Control (No Intervention): Exercice Session without any music

INTERVENTIONS:
Other: Music listening during physical exercise — Exposure to music played at different phases of the physical activity
  Arms: MFH; MSH; MT

SUMMARY:
Affective phenomena, such as core affect, remembered pleasure, or forecasted pleasure, play a key role in promoting physical activity (PA) behaviour, especially among inpatients. The use of music has been shown to be a particularly cost-effective and low-friction approach to promoting positive affective valence during PA. However, interventions using music to improve exercise-related affective phenomena among inpatients are lacking. This study will aim to investigate an intervention that combines the effects of music with the "peak-end rule" on core affective responses (valence and arousal), remembered pleasure, and forecasted pleasure associated with exercise sessions among cardiac rehabilitation inpatients.

The primary objective of the present study will be to examine the effect of differentiated music exposure on core affective responses, ratings of perceived exertion and psychophysiological responses to moderate-intensity continuous training (MICT), as well as on associated remembered pleasure, exercise enjoyment, and forecasted pleasure. A secondary objective will be to assess the potential mediating effect of affective valence at the end of the MICT on remembered pleasure and exercise enjoyment. A third objective will be to assess the effect of MICT with or without music on an emotional rating task, together with pupillometric measures. Finally, the study will examine the influence of remembered pleasure on subsequent forecasted pleasure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in an inpatient 3-week cardiac exercise-based rehabilitation programme
* Age range 50-75 years
* Can withstand the study protocol without undue risk
* Able to provide written consent

Exclusion Criteria:

* Contraindication to physical activity in view of the health status
* Presence of cognitive or psychological disorder
* Hearing impairment with or without hearing aids

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Affective valence during the moderate intensity continuous training | 22 minutes
  Mesured with filling scale (FS)

SECONDARY OUTCOMES:
Affective arousal during the moderate-intensity continuous training | 25 minutes
  Affective arousal will be measured at five time points ( Minute 3, Minute 12, Minute 13, Minute 22, and Minute 25) using the Felt Arousal Scale (Svebak & Murgatroyd, 1985), a single-item bipolar rating scale using the sentence "How aroused do you actually feel?" with possible responses ranging from 1 (low arousal) to 6 (high arousal).
Rating of perceived exertion during the moderate-intensity continuous training | 5 minutes after each training session
  Remembered pleasure will be measured 5 min after each training session using a visual analogy scale presented on a Samsung Galaxy Tab ranging from -100 (very unpleasant) to +100 (very pleasant) in intervals of 1 (Zenko et al., 2016). Participants will be asked to answer the following question: "How did the exercise session make you feel?" (Hutchinson et al., 2023).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided